CLINICAL TRIAL: NCT02786953
Title: Sleep Coach: Sleep Promotion to Improve Diabetes Management in Adolescents With T1D
Brief Title: Sleep Promotion to Improve Diabetes Management in Adolescents With T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Jaser, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151271
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Sleep; Adherence; Diabetes Management; Adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Promotion (Experimental): Behavioral sleep-promoting intervention, including components such as limiting caffeine, establishing a media curfew, and positive bedtime routines, as well as needs unique to adolescents with T1D, such as fear of hypoglycemia.
  Interventions: Behavioral: Sleep Promotion
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Sleep Promotion — Behavioral intervention to improve sleep quality and duration.
  Arms: Sleep Promotion

SUMMARY:
Adolescents with type 1 diabetes (T1D) are at increased risk for problems with adherence and suboptimal glycemic control, and novel approaches are needed to improve outcomes in this high-risk population. The majority of adolescents obtain insufficient sleep (defined as <8 hours/night), and sleep disturbance has been significantly associated with poorer adherence and predicted greater problems with quality of life and worse glycemic control. Yet, no interventions have addressed sleep in youth with T1D. Working from a biopsychosocial and contextual model of sleep, the investigators propose to tailor a sleep-promoting intervention to meet the needs of adolescents with T1D by conducting interviews with to identify the barriers and facilitators to adequate sleep specific to this population. The sleep-promoting intervention will be developed and tested, building on successful sleep interventions in other populations, including components such as limiting caffeine, establishing a media curfew, and positive bedtime routines, while addressing the needs unique to adolescents with T1D, such as fear of hypoglycemia. The study will be conducted by a multidisciplinary team, consisting of Sarah Jaser, PhD, a pediatric psychologist, and two co-investigators, Beth Malow, MD, MS, a neurologist with specialty in sleep medicine, and Jill Simmons, MD, a pediatric endocrinologist. Sleep is a potentially modifiable risk factor that may have both a physiological and behavioral impact on diabetes outcomes. Given the strong associations between sleep and diabetes outcomes in the preliminary data, and recent evidence from sleep restriction studies indicating the impact of insufficient sleep on insulin sensitivity, behavior, and mood, there is reason to believe that a sleep-promoting intervention has the potential to improve outcomes in adolescents with T1D indirectly by improving adherence and directly through its effect on metabolic function. Therefore, the proposed study offers a novel approach to improve adherence, quality of life, and glycemic control in adolescents with T1D.

DETAILED DESCRIPTION:
Working from a biopsychosocial and contextual model of sleep, this study will pilot test a sleep-promoting intervention tailored to meet the needs of adolescents with T1D, building on successful sleep interventions in other populations, including components such as limiting caffeine, establishing a media curfew, and positive bedtime routines, while addressing the needs unique to adolescents with T1D, such as fear of hypoglycemia. The study will be conducted by a multidisciplinary team, consisting of Sarah Jaser, PhD, a pediatric psychologist, and two co-investigators, Beth Malow, MD, MS, a neurologist with specialty in sleep medicine, and Jill Simmons, MD, a pediatric endocrinologist. Sleep is a potentially modifiable risk factor that may have both a physiological and behavioral impact on diabetes outcomes. Given the strong associations between sleep and diabetes outcomes in the preliminary data, and recent evidence from sleep restriction studies indicating the impact of insufficient sleep on insulin sensitivity, behavior, and mood, there is reason to believe that a sleep-promoting intervention has the potential to improve outcomes in adolescents with T1D indirectly by improving adherence and directly through its effect on metabolic function. Therefore, the proposed study offers a novel approach to improve adherence, quality of life, and glycemic control in adolescents with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes for at least 12 months
* Speak and read English
* Report Insufficient sleep (< 8 hours/night most school nights)

Exclusion Criteria:

* Other major health problems or sleep disorders (other than insomnia)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2019-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Jaser, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant consented, completed baseline data, then withdrew
Period: Overall Study
Arm/Group | Sleep Promotion | Usual Care
Started | 20 | 19
Baseline Teen Survey Data Completed | 20 | 18 (One participant withdrawn and data excluded due to becoming ineligible due to a new diagnosis)
Baseline Parent Survey Completed | 20 | 18 (One participant withdrawn and data excluded due to becoming ineligible due to a new diagnosis)
Actigraph Data Complete | 14 | 17 (One participant withdrawn and data excluded due to becoming ineligible due to a new diagnosis)
A1C Data Baseline | 20 | 18 (One participant withdrawn and data excluded due to becoming ineligible due to a new diagnosis)
Session 1 Completed | 17 | 0
Session 2 Completed | 16 | 0
Session 3 Completed | 16 | 0
3 Month Teen Survey Completed | 17 | 18
3 Month Parent Survey Completed | 17 | 18
A1C 3 Month | 15 | 17
Completed | 17 | 18
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 family enrolled and was randomized to usual care. Teen was diagnosed with a condition that caused them to be excluded, so they were removed from baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Promotion | Usual Care | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.85 (1.27) | 15.72 (1.32) | 15.26 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 15 | 14 | 29
  Non-White | 4 | 2 | 6
  Hispanic | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38
Annual Income [Count of Participants; unit: Participants]
  <$39,999 | 7 | 2 | 9
  $40,000-$79,999 | 7 | 5 | 12
  >$80,000 | 5 | 10 | 15
  Missing | 1 | 1 | 2
Treatment Type [Count of Participants; unit: Participants]
  Insulin Pump | 12 | 11 | 23
  Injection | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality: Baseline
Description: Sleep quality will be measured with the Pittsburgh Sleep Quality Index total score. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 20 | 18
score on a scale | 4.3 (1.7) | 4.5 (1.5)

2. Primary Outcome: Sleep Quality 3 Months
Description: as for outcome 1
Time Frame: 3 months
Population: includes only participants with baseline and 3 month data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 17 | 18
score on a scale | 3.9 (1.5) | 4.8 (1.6)

3. Primary Outcome: Glycemic Control (HbA1c) Baseline
Description: HbA1C is a measure of average blood glucose levels. It is measured quarterly at regular clinic visits.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of glycosylated Hgb
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 20 | 18
percentage of glycosylated Hgb | 9.4 (2.2) | 9.1 (1.5)

4. Primary Outcome: Glycemic Control (HbA1c) 3 or 6 Months
Description: HbA1C is a measure of average blood glucose levels. It is measured quarterly at regular clinic visits.
Time Frame: 3 months or 6 months
Population: Some participants missed the 3 month appointment, so the final result is a combination of 3 month and 6 month values
Measure: Mean (Standard Deviation); unit: percentage of glycosylated Hemoglobin
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 17 | 17
percentage of glycosylated Hemoglobin | 9.2 (2.0) | 9.2 (1.2)

5. Primary Outcome: Sleep Duration: Baseline
Description: Sleep duration will be measured with actigraphy (total sleep time)
Time Frame: baseline
Population: only participants with usable actigraph data
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 14 | 17
hours | 6.85 (0.82) | 6.69 (1.00)

6. Primary Outcome: Sleep Duration: 3 Months
Description: Sleep duration will be measured with actigraphy (total sleep time)
Time Frame: 3 months
Population: only participants with usable actigraph data
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 13 | 12
hours | 7.02 (0.78) | 6.37 (0.92)

7. Secondary Outcome: Quality of Life (PedsQL)
Description: The PedsQL, Type 1 Diabetes module, a self-report measure of quality of life will be used. Scaled scores range from 0-100, and higher scores indicate better quality of life.
Time Frame: Baseline and 3 months
Population: only participants with both baseline and 3 month data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 17 | 18
score on a scale
  baseline | 70.3 (8.0) | 74.5 (8.6)
  3 months | 72.5 (10.3) | 75.4 (9.9)

8. Secondary Outcome: Adherence (Self Care Inventory) Parent
Description: The parent versions of the Self Care Inventory will be used to measure adherence to the diabetes treatment regimen. Mean scores are calculated, ranging from 1-5, with higher scores indicating better adherence.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 17 | 18
score on a scale
  baseline | 3.7 (.66) | 3.8 (.69)
  3 months | 3.8 (.84) | 3.7 (.73)

9. Secondary Outcome: Adherence (Self Care Inventory) Teen
Description: The teen versions of the Self Care Inventory will be used to measure adherence to the diabetes treatment regimen. Mean scores are calculated, ranging from 1-5, with higher scores indicating better adherence.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Promotion | Usual Care
Number analyzed (Participants) | 17 | 18
score on a scale
  baseline | 3.9 (.76) | 3.7 (.79)
  3 months | 3.8 (.46) | 3.9 (.59)

ADVERSE EVENTS:
Time Frame: baseline to 3 months
Arm/Group | Sleep Promotion | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
pilot study with small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT02786953/Prot_SAP_000.pdf